CLINICAL TRIAL: NCT05117034
Title: Pre-emptive Intravenous Morphine for Acute Post-craniotomy Pain: a Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: Pre-emptive Intravenous Morphine for Acute Post-craniotomy Pain.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Barak Cohen, MD, Vice chair, department of Anesthesia, Intensive Care, and Pain Management, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0193-21-TLV-OG
Record Dates: First submitted 2021-11-02; First posted 2021-11-11 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Pain, Postoperative; Anesthesia; Analgesia
Keywords: Craniotomy; Post-craniotomy pain; Opioid analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Morphine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A double-blind randomized controlled trial. Participating adults having craniotomy surgery will be randomized in a 1:1 ratio to intraoperative intravenous administration of 0.08 mg/kg morphine at dura closure, or a matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morphine (Experimental): Intraoperative intravenous administration of 0.08 mg/kg morphine at dura closure.
  Interventions: Drug: Morphine
- Placebo (Placebo Comparator): Intraoperative intravenous administration of 0.08 ml/kg NaCl 0.9% at dura closure.
  Interventions: Drug: Nacl 0.9%

INTERVENTIONS:
Drug: Morphine — Intraoperative intravenous administration of 0.08 mg/kg morphine at dura closure.
  Arms: Morphine
Drug: Nacl 0.9% — Intraoperative intravenous administration of 0.08 ml/kg NaCl 0.9% at dura closure.
  Arms: Placebo

SUMMARY:
We propose a double-blind randomized controlled trial to evaluate the effect of intravenously administered morphine at surgery conclusion on acute postoperative pain in patients recovering from craniotomy surgery. Participating adults having craniotomy surgery will be randomized in a 1:1 ratio to intraoperative intravenous administration of 0.08 mg/kg morphine at dura closure, or a matching placebo.

DETAILED DESCRIPTION:
After confirming eligibility, patients will be approached by one of the study researchers for potential participation. After a thorough explanation, written informed consent will be obtained.

General anesthesia will be induced with propofol (2-3 mg/kg), and either remifentanil (1 mcg/kg) or fentanyl (2 mcg/kg). Lidocaine (1 mg/kg) and rocuronium (0.6 mg/kg) will be allowed and left to the discretion of the caregivers. Anesthesia will be maintained with infusions of propofol and remifentanil, and titrated to maintain hemodynamic goals and evaluation of anesthesia depth by somatosensory or motor evoked potentials according to clinical requirements. Ketamine and fentanyl administration will not be allowed at the maintenance phase. No additional IV opioids will be allowed during surgery. Other analgesics such as dipyrone and non-steroidal anti-inflammatory agents (such as diclofenac) will not be allowed during surgery or during PACU stay. At dura closure, patients will be randomized by a web-based randomization service in a 1:1 ratio. The intervention group will receive 0.08 mg/kg intravenous morphine (0.08 ml/kg), while the control group will receive 0.08 ml/kg 0.9% NaCl. The research solution (morphine/0.9% NaCl) will be administered via IV infusion over ten minutes. Randomization and study drug preparation will be performed by a research team-member, uninvolved in data collection, analysis, or patient care.

Both groups will receive acetaminophen (1 gr) at dura closure. Steroids and other anti-emetic medications will be allowed. Remifentanyl and propofol infusions will be discontinued at the end of the surgery during wound dressing. All patients will have orders for intravenous morphine administration in PACU for breakthrough pain as acceptable and according to the orders prescribed by anesthesiologist assigned for the case/the attending anesthesiologist in PACU. The research team/protocol does not interfere with morphine administration during PACU stay. All caregivers will be blinded to treatment allocation.

Patient's monitoring at the operating room and during transportation to the PACU will be done by the anesthesiologist assigned for the case. Patient's monitoring during PACU stay will be done by the PACU team and according to the patient's clinical status according to PACU protocol. Patients will be followed during PACU stay by a study team member blinded to the treatment allocation. The study team member will measure and record pain score (NRS), sedation score (Ramsay score) and PONV at admission to PACU and 30 minutes after admission to PACU. The research team, according the research hypothesis is interested in measuring pain (via NRS) while the patient is fully conscious and alert. Additional data regarding the surgery, anesthesia, recovering from anesthesia and PACU stay will be collected retroactively from computer system data (metavision, chameleon).

Demographic and clinical data will be collected on the day of surgery. Surgical and anesthetic data, laboratory results, details regarding side effects, time of first morphine requirement, total morphine consumption in PACU, and pain scores (NRS) at POD1 and POD2 will be collected from computerized patient files.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Scheduled for elective craniotomy for resection of supra-tentorial intracranial tumor that requires cranium sawing, dural opening and excision of tumor, under general anesthesia.
* Age 18 - 80 years.
* American Society of Anesthesiologists' physical status I-III.
* Body mass index (BMI) under 35 kg/m2.

Exclusion Criteria:

* Pregnant or current breastfeeding patients.
* Patients unable to provide informed consent or in need of a legal authorized representative.
* Patients with neurological disorders preventing a good understanding of the pain numerical reporting scale (NRS) before surgery.
* Patients with pre-operative aphasia.
* Patients with chronic pain or chronic use of opioids.
* Patients with current alcohol or drug abuse.
* Expected delayed extubation.
* Patients with documented allergy to opioids or acetaminophen.
* Preoperative Glasgow Coma Scale <15.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
First NRS pain score. | Up to 1 hour from PACU admission
  The numeric rating scale (NRS), a validated tool used to assess patients' self-reported pain level, will be taken at admission to the post anesthesia care unit (PACU). NRS score ranges from 0 to 10, with higher scores representing worse pain.

SECONDARY OUTCOMES:
Time to first rescue morphine administration | During 2 hours from PACU admission.
  Time measured (in minutes) from admission to the post anesthesia care unit (PACU) to patient's first rescue morphine administration.
Total morphine consumption | During 2 hours from PACU admission.
  Total dosage of rescue morphine given to the patient during the first two hours of PACU stay.

OTHER OUTCOMES:
Systolic and mean arterial pressure. | During 30 minutes from PACU admission.
  Systolic and mean arterial pressure measured on admission to PACU and 30 minutes after admission to PACU.
Time-weighted average NRS pain score during the first two postoperative days. | During 48 hours from PACU admission.
  The sum of the portion of each time period (measured in hours) for specific NRS value multiplied by the specific NRS score during the time period divided by 48 hours.
NRS pain score 30 minutes after admission to PACU. | During 30 minutes from PACU admission.
  The numeric rating scale (NRS), a validated tool used to assess patients' self-reported pain level, will be taken 30 minutes after admission to the post anesthesia care unit (PACU). NRS score ranges from 0 to 10, with higher scores representing worse pain.
Sedation level. | During 30 minutes from PACU admission.
  Sedation level as measured by the Ramsay Agitation and Sedation Scale (RASS) score on admission to PACU and 30 minutes after PACU admission.
Arterial CO2 partial pressure (PaCO2). | During 2 hours from PACU admission.
  Arterial CO2 partial pressure (PaCO2) on PACU admission.
Postoperative nausea or vomiting. | During 2 hours from PACU admission.
  Postoperative nausea or vomiting, as captured by patients' response to the question "are you feeling nauseated?" or a document event of vomiting during the first two hours of PACU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Or Goren, MD, Principal Investigator — Department of Anesthesia, Intensive Care, and Pain Management, Tel-Aviv Medical Center
Locations (1):
- Tel-Aviv Medical Center, Sackler faculty of medicine, Tel-Aviv University, Israel, Tel Aviv, Israel